CLINICAL TRIAL: NCT04249011
Title: Assessment of Sleep-related Respiratory Disorders at High Altitude With the WatchPAT200TMU Compared to PSG.
Brief Title: WatchPAT Compared to PSG at 8500'
Status: Completed | Type: Observational
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: WP200U-Altitude-001
Record Dates: First submitted 2020-01-20; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Sleep Disorder; Breathing-Related
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subjects who consent to participate in the research will undergo a simultaneous recording of inlab PSG and WatchPAT200 for comparing the WatchPAT data to PSG at an altitude of 8500'.

DETAILED DESCRIPTION:
The efficacy of the WP200U will be evaluated by comparing it to the PSG manual scoring of sleep disordered breathing (SDB) parameter using the PSG manual scoring as a "gold standard"

ELIGIBILITY:
Inclusion Criteria:

* Male and females ≥ age 17yrs
* Subject is able to read understand and sign the informed consent form.
* Willing to sleep with the WP200U and PSG simultaneously in the sleep lab.

Exclusion Criteria:

* Use of one of the following medications: alpha blockers, short acting nitrates (less than 3 hours before the study).

  * Any condition that in the opinion of the investigator may adversely affect the safety of the patient or would limit the patient ability to complete the study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects referred to a sleep lab for full PSG.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Comparison of AHI and ODI as scored automatically by the WatchPAT compared to manual scoring of full night PSG. | 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: Koby Sheffy, Phd, Study Director — Itamar-Medical, Israel
Locations (1):
- Mountain Sleep Diagnostics, Woodland Park, Colorado, United States